CLINICAL TRIAL: NCT04875195
Title: A Phase 2 Study of Pembrolizumab (MK-3475) Every 6 Weeks (Q6W) in Participants With Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL) or Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL)
Brief Title: A Study of Pembrolizumab (MK-3475) in Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL) or Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) (MK-3475-B68)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-B68; MK-3475-B68 (Other: MSD); 2024-510979-38-00 (Registry Identifier: EU CT); U1111-1302-8634 (Registry Identifier: UTN); 2020-005609-20 (EudraCT Number)
Record Dates: First submitted 2021-04-27; First posted 2021-05-06 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Hodgkin's Lymphoma; Primary Mediastinal Large B-cell Lymphoma (PMBCL)
Keywords: PD1; PD-1; PDL1; PD-L1
MeSH Terms: conditions — Hodgkin Disease | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Pembrolizumab (MK-3475), 400 mg, Q6W, intravenous (IV) infusion, Day 1 then Q6W up to 18 doses.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab, 400 mg, Q6W, intravenous (IV) infusion.
  Other Names: MK-3475; SCH 900475; KEYTRUDA®

SUMMARY:
The primary objective of the study is to evaluate the objective response rate (ORR), by cohort, rrcHL and rrPMBCL, as assessed by the investigator according to Lugano classification criteria 2014 in participants treated with pembrolizumab every six weeks (Q6W).

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of cHL or PMBCL, according to the World Health Organization (WHO) classification [Swerdlow, S. H., et al 2008].
* Has radiographically measurable cHL or PMBCL disease as per Lugano classification with at least 1 nodal lesion (which has not been previously radiated) that is >15 mm in long axis, regardless of the length of the short axis, and/or extranodal lesion of >10 mm in long and short axis.

PMBCL-Specific Disease Characteristics:

* Have relapsed or refractory PMBCL and:
* Have relapsed after auto-stem cell transplant (SCT) or have failed to achieve a CR or PR within 60 days of auto-SCT. Participants may have received intervening therapy after auto-SCT for relapsed or refractory disease, in which case they must have relapsed after or be refractory to their last treatment.

OR

- For participants who are ineligible for auto-SCT, have received at least ≥2 lines of prior therapy and have failed to respond to or relapsed after their last line of treatment. At least 1 of the prior lines of therapy must contain a rituximab-based regimen.

Note: Participants should not need urgent cytoreductive therapy.

* Relapsed Disease: disease progression after achieving an overall response of PR or CR in response to the most recent therapy
* Refractory Disease: failure to achieve CR or PR to the most recent therapy.

cHL-Specific Disease Characteristics:

* Have relapsed or refractory cHL and:
* Have relapsed during their last cHL regimen after receiving at least 2 cycles of therapy or within 12 months after completing the last regimen for cHL.

OR

* Have received at least ≥1 line of prior multiagent therapy with/without brentuximab vedotin (excluding radiation) or auto-SCT for cHL and have failed to respond to or relapsed after their last line of treatment.

  * Relapsed Disease: disease progression after achieving an overall response of PR or CR to the most recent therapy.
  * Refractory Disease: failure to achieve CR or PR to the most recent therapy.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
* Is not a woman of child bearing potential (WOCBP). OR
* Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), for at least 120 days after the last dose of study intervention.
* Submit an evaluable core lymph node biopsy for biomarker analysis from an archival (>60 days) or newly obtained (within 30 days) core or incisional biopsy at Screening which was not previously irradiated. Note: If no archival tissue is available, 2 new fresh core needle samples are required.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Life expectancy >3 months.
* Adequate organ function.

Exclusion Criteria:

* Has undergone solid organ transplant at any time, or prior allogeneic hematopoietic SCT within the last 5 years
* Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), or serious cardiac arrhythmia requiring medication
* Has pericardial effusion or clinically significant pleural effusion
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers
* Is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) <3 days prior to the first dose of study intervention. Note: Participants who receive daily steroid replacement therapy are an exception
* Has received prior monoclonal antibody within 4 weeks prior to first dose of study intervention or has not recovered (i.e., ≤Grade 1 or at baseline) from adverse event (AEs) due to agents administered more than 4 weeks earlier
* Has received prior therapy with an anti-programmed cell death 1 protein (PD-1), anti-programmed cell death ligand 1 (PD-L1), or anti-programmed cell death ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137)
* Has received prior chimeric antigen receptor T-cell (CAR-T) therapy
* Has received prior systemic anticancer therapy, or radiotherapy, including investigational agents within 4 weeks prior to the first dose of study intervention. Note: If the participant had a major operation, the participant must have recovered adequately from the procedure and/or any complications from the operation before starting study intervention
* Has received prior radiotherapy within 2 weeks of start of study intervention or have had a history of radiation pneumonitis. Participants must have recovered from all radiation-related toxicities, and not require corticosteroids
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study drug
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Has known active central nervous system (CNS) lymphoma involvement or active CNS involvement by lymphoma
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority
* Has a known history of Hepatitis B (defined as hepatitis B surface antigen (HBsAg) reactive) or known active Hepatitis C virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2025-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (27):
- United States (3):
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA-Hematology and Medical Oncology ( Site, Torrance, California
  - Tulane Medical Center ( Site 0110), New Orleans, Louisiana
  - Anne Arundel Medical Center-Anne Arundel Oncology and Hematology ( Site 0125), Annapolis, Maryland
- Brazil (2):
  - Hospital Erasto Gaertner ( Site 1703), Curitiba, Paraná
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 1701), Barretos, São Paulo
- Cross Cancer Institute ( Site 0207), Edmonton, Alberta, Canada
- Czechia (3):
  - Fakultni nemocnice Brno Bohunice-Interni hematologicka a onkologicka klinika ( Site 0302), Brno, Brno-mesto
  - Fakultni nemocnice Kralovske Vinohrady-Interni hematologicka klinika ( Site 0303), Prague, Praha 10
  - Fakultni nemocnice Hradec Kralove-IV. interni hematologicka klinika ( Site 0304), Hradec Králové
- France (2):
  - Centre Hospitalier Universitaire Dijon Bourgogne - Hôpital François Mitterrand ( Site 0401), Dijon, Cote-d Or
  - Gustave Roussy ( Site 0402), Villejuif, Île-de-France Region
- Italy (3):
  - Fondazione IRCCS Policlinico San Matteo ( Site 0509), Pavia, Lombardy
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO-EMATOLOGIA I ( Site 0507), Palermo, Sicily
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 0503), Napoli
- Poland (3):
  - Szpital Kliniczny im. Przemienienia Panskiego Uniwersytetu M-Oddzial Hematologii i Transplantacji S, Poznan, Greater Poland Voivodeship
  - Pratia MCM Krakow ( Site 0064), Krakow, Lesser Poland Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Hematologii i Transplantologii ( Site 0063), Gdansk, Pomeranian Voivodeship
- Russia (3):
  - The National Medico-Surgical Center N.I. Pirogov ( Site 0801), Moscow, Moscow
  - Moscow City Clinical Hospital S.P. Botkin ( Site 0803), Moscow, Moscow
  - Almazov National Medical Research Centre ( Site 0807), Saint Petersburg, Sankt-Peterburg
- South Africa (3):
  - Netcare Pretoria East Hospital-Albert Alberts Stem Cell Transplant Centre ( Site 0902), Centurion, Gauteng
  - Wits Clinical Research ( Site 0904), Johannesburg, Gauteng
  - Groote Schuur Hospital ( Site 0906), Cape Town, Western Cape
- Turkey (Türkiye) (2):
  - Ege University Medicine of Faculty ( Site 1105), Bornova, İzmir
  - Ankara University Department of Hematology, Clinical Research Unit ( Site 1101), Ankara
- Ukraine (2):
  - CNPE Regional Center of Oncology ( Site 1305), Kharkiv, Kharkivs’ka Oblast’
  - National Cancer Institute ( Site 1303), Kyiv, Kyivska Oblast

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26325&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL): Participants with rrcHL received pembrolizumab 400 mg as an intravenous (IV) infusion on Day 1, then every six weeks (Q6W) up to 18 doses.
- Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL): Participants with rrPMBCL received pembrolizumab 400 mg as an intravenous (IV) infusion on Day 1, then every six weeks (Q6W) up to 18 doses.
Period: Overall Study
Arm/Group | Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL) | Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL)
Started | 60 | 6
Completed | 0 | 0
Not Completed | 60 | 6
Not completed — Death | 9 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Ongoing in study | 49 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL) | Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) | Total
Number analyzed (Participants) | 60 | 6 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (16.1) | 32.5 (8.6) | 37.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 4 | 35
  Male | 29 | 2 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 0 | 6
  Not Hispanic or Latino | 50 | 6 | 56
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 49 | 5 | 54
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Lugano Classification as Assessed by Investigator
Description: ORR was defined as the percentage of the participants who had complete response (CR) or partial response (PR) and was evaluated using computed tomography (CT) and metabolic imaging (fluorodeoxyglucose- positron emission tomography (FDG-PET)). CR is complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). The percentage of participants treated with pembrolizumab Q6W, by cohort, rrcHL and rrPMBCL, who experienced CR or PR as assessed by investigator is presented.
Time Frame: Up to approximately 30 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL) | Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL)
Number analyzed (Participants) | 60 | 6
Percentage of Participants | 66.7 [53.3 to 78.3] | 50.0 [11.8 to 88.2]

2. Secondary Outcome: ORR Per Lugano Classification as Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of the participants who had complete response (CR) or partial response (PR) and was evaluated using computed tomography (CT) and metabolic imaging (fluorodeoxyglucose-positron emission tomography (FDG-PET)). CR is complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). The percentage of participants treated with pembrolizumab Q6W, by cohort, rrcHL and rrPMBCL, who experienced CR or PR as assessed by BICR is presented.
Time Frame: Up to approximately 30 months
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL) | Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL)
Number analyzed (Participants) | 60 | 6
Percentage of Participants | 70.0 [56.8 to 81.2] | 66.7 [22.3 to 95.7]

3. Secondary Outcome: Duration of Response (DOR) Per Lugano Classification as Assessed by Investigator
Description: For participants who demonstrate a CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. Participants will be evaluated using CT and metabolic imaging (FDG-PET). CR is complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). DOR as assessed by investigator is presented among participants who demonstrated CR or PR.
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: DOR Per Lugano Classification as Assessed by BICR
Description: For participants who demonstrate a CR or PR, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. Participants will be evaluated using CT and metabolic imaging (FDG-PET). CR is complete metabolic (no/minimal FDG uptake) and radiologic response (target lesions regress to ≤1.5 cm in longest transverse diameter of a lesion) and no new lesions. PR is partial metabolic (moderate/high FDG uptake) and radiologic response (≥50% decrease in sum of product diameters for multiple lesions of up to 6 target measurable nodes and extranodal sites, no increase in lesions, and spleen regressed by >50% in length beyond normal). DOR as assessed by BICR is presented among participants who demonstrated CR or PR.
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Area Under the Curve (AUC) Early Cycle of Pembrolizumab
Description: AUC was defined as a measure of pembrolizumab exposure that was calculated as the product of serum drug concentration and time. Blood samples were collected to determine the AUC of pembrolizumab during Cycle 1 (early cycle). A cycle was 6 weeks.
Time Frame: Predose on Day 1 and Day 42 of Cycle 1 (cycle length=6 weeks)
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment. The analysis was pre-specified to be a pooled analysis of all participants rrcHL or rrPMBCL.
Measure: Geometric Mean (95% Confidence Interval); unit: day*µg/mL
Groups:
- rrcHL or rrPMBCL: Participants with rrcHL or rrPMBCL received pembrolizumab 400 mg as an intravenous (IV) infusion on Day 1, then every six weeks (Q6W) up to 18 doses.
Arm/Group | rrcHL or rrPMBCL
Number analyzed (Participants) | 66
day*µg/mL | NA [NA to NA] — AUC was determined by trapezoidal methods using interpolation between data points. Thus, at least 3 data points in the terminal phase excluding Tmax (i.e., end of infusion) were required to determine AUC. Due to sparse PK sampling schedule, per participant data could not be calculated.

6. Secondary Outcome: Area Under the Curve (AUC) Steady State of Pembrolizumab
Description: AUC was defined as a measure of pembrolizumab exposure that was calculated as the product of serum drug concentration and time. Blood samples were collected to determine the AUC of pembrolizumab during Cycle 4 (steady state). A cycle was 6 weeks.
Time Frame: Predose on Day 1 and Day 42 of Cycle 4 (cycle length=6 weeks)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: day*µg/mL
Arm/Group | rrcHL or rrPMBCL
Number analyzed (Participants) | 66
day*µg/mL | NA [NA to NA] — AUC was determined by trapezoidal methods using interpolation between data points. Thus, at least 3 data points in the terminal phase excluding Tmax (i.e., end of infusion) were required to determine AUC. Due to sparse PK sampling schedule, per participant data could not be calculated.

7. Secondary Outcome: Maximum Serum Concentration (Cmax) Early Cycle of Pembrolizumab
Description: Cmax is defined as the maximum serum drug concentration. Blood samples were collected to determine the Cmax of pembrolizumab during Cycle 1 (early cycle).
Time Frame: Predose on Day 1 of Cycle 1 and end of infusion on Day 1 of Cycle 1 (cycle length = 6 weeks)
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment and had Cycle 1 end of infusion concentration available. A cycle is 6 weeks. The analysis was pre-specified to be a pooled analysis of all participants rrcHL or rrPMBCL.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | rrcHL or rrPMBCL
Number analyzed (Participants) | 61
μg/ml | 127.5 [120.0 to 135.4]

8. Secondary Outcome: Maximum Serum Concentration (Cmax) Steady State of Pembrolizumab
Description: Cmax is defined as the maximum serum drug concentration. Blood samples were collected to determine the Cmax of pembrolizumab during Cycle 4 (steady state).
Time Frame: Predose on Day 1 of Cycle 4, and end of infusion on Day 1 of Cycle 4 (cycle length = 6 weeks)
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment and had Cycle 4 end of infusion concentration available. A cycle is 6 weeks. The analysis was pre-specified to be a pooled analysis of all participants rrcHL or rrPMBCL.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | rrcHL or rrPMBCL
Number analyzed (Participants) | 41
μg/ml | 154.8 [141.5 to 169.4]

9. Secondary Outcome: Trough Serum Concentration (Ctrough) Early Cycle of Pembrolizumab
Description: Ctrough is defined as the lowest serum drug concentration. Blood samples were collected to determine the Ctrough of pembrolizumab during Cycle 1 (early cycle).
Time Frame: Predose on Day 1 of Cycle 1 and Day 42 of Cycle 1 (cycle length = 6 weeks)
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment and had Cycle 1 trough concentration available. A cycle is 6 weeks. The analysis was pre-specified to be a pooled analysis of all participants with rrcHL or rrPMBCL.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | rrcHL or rrPMBCL
Number analyzed (Participants) | 61
μg/ml | 17.9 [16.3 to 19.7]

10. Secondary Outcome: Trough Serum Concentration (Ctrough) Steady State of Pembrolizumab
Description: Ctrough is defined as the lowest serum drug concentration. Blood samples were collected to determine the Ctrough of pembrolizumab during Cycle 4 (steady state).
Time Frame: Predose on Day 1 of Cycle 1 and Day 42 of Cycle 4 (cycle length = 6 weeks)
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment and had Cycle 4 trough concentration available. A cycle is 6 weeks. The analysis was pre-specified to be a pooled analysis of all participants with rrcHL or rrPMBCL.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/ml
Arm/Group | rrcHL or rrPMBCL
Number analyzed (Participants) | 44
μg/ml | 33.8 [29.9 to 38.4]

11. Secondary Outcome: Antidrug Antibody Levels (ADA) for Pembrolizumab
Description: Blood samples were collected and assayed for anti-pembrolizumab antibodies presence using a validated electrochemiluminescence immunoassay. Negative ADA refers to all pre-treatment and postdose samples negative in the assay for antibodies against pembrolizumab and the concentration of pembrolizumab in the last postdose sample below the drug tolerance level. Treatment emergent positive was defined as pre-treatment sample negative and at least one postdose sample positive in the assay or pre-treatment and postdose sample positive with an increase in titer (≥2 fold of baseline). Non-treatment emergent positive was defined as pre-treatment sample positive and postdose sample negative or pre-treatment and postdose sample positive with a postdose titer <2 fold of baseline. Neutralizing positive was defined as at least 1 of the ADA positive samples test positive in the neutralizing assay.
Time Frame: Predose 0-4 hours on Cycle1 Day1, Cycle2 Day1, Cycle4 Day1, Cycle5 Day1, Cycle7 Day1, Cycle9 Day1, Cycle13 Day1, Cycle17 Day1 and end of infusion on Cycle1 Day1, Cycle4 Day1 and anytime on Cycle1 Day22 and Cycle4 Day22 (cycle length = 6 weeks)
Population: The analysis population consisted of all participants who received ≥1 dose of study treatment and had a negative ADA or positive ADA status. The analysis was pre-specified to be a pooled analysis of all participants with rrcHL or rrPMBCL.
Measure: Count of Participants; unit: Participants
Arm/Group | rrcHL or rrPMBCL
Number analyzed (Participants) | 64
Participants
  Negative | 62
  Treatment emergent positive | 1
  Non-Treatment emergent positive | 1
  Neutralizing positive | 0

12. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2026-12

13. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to AE
Description: as for outcome 12
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: Up to approximately 30 months
Description: The analysis population for AEs included all participants who received ≥1 dose of study treatment. MedDRA preferred terms "neoplasm progression (NP)", "malignant NP" and "disease progression" not related to study treatment are excluded.
Arm/Group | Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL) | Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL)
All-Cause Mortality (participants affected / at risk) | 9/60 | 3/6
Serious Adverse Events (participants affected / at risk) | 5/60 | 0/6
Other Adverse Events (participants affected / at risk) | 38/60 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL) (N=60) | Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastric stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed or Refractory Classical Hodgkin's Lymphoma (rrcHL) (N=60) | Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) (N=6)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 1 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 8 (8) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 1 (3)
COVID-19 (Infections and infestations) | 13 (13) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 4 (7) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (18) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 5 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (8) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Anhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT04875195/Prot_SAP_000.pdf